CLINICAL TRIAL: NCT01830998
Title: Study of Cognitive Dysfunction and Diabetes
Brief Title: Early Detection of Cognitive Dysfunction in Diabetes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wuhan General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, zhipeng xu, doctor, Wuhan General Hospital of Guangzhou Military Command
Other Study IDs: 20130401
Record Dates: First submitted 2013-04-01; First posted 2013-04-12 (Estimated); Last update posted 2014-12-10 (Estimated); Status verified 2014-12

CONDITIONS: Dementia; DM; MCI
Keywords: Dementia; Olfactory
MeSH Terms: conditions — Dementia; Anosmia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: None Retained — serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- control,MCI, Olfactory dsfunction: There are different groups:control,MCI, Olfactory dsfunction.
- control, MCI: control and MCI group.Glycaemic control
- control and MCI: treatment and without treatment
- MCI and Olfactory function: observation between MCI and Olfactory function groups.

SUMMARY:
The rate of cognitive decline due to ageing is increased 1.5-fold to 2.0-fold in individuals with type 2 diabetes.There are no established specific treatment measures to prevent or ameliorate cognitive impairments in patients with diabetes. we want to detecte early clinical dementia in diabete.

DETAILED DESCRIPTION:
Clinically relevant cognitive decrements in relation to diabetes mainly occur during two crucial periods in life: the period of brain development in childhood, and the period when the brain undergoes neurodegenerative changes associated with ageing.Potential leads for treatment are to optimise glycaemic control and avoid and treat vascular risk factors.we want to detecte early clinical dementia in diabete by MMSE and Olfactory function.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 2 diabetes(Age>50 years)

Exclusion Criteria:

* with stroke or other complications.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2012-01; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
MMSE Olfactory function dementia | 2 years
  MMSE,Olfactory function and PET(fMRI) were observed.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Wuhan general hospital of Guangzhou Command, Wuhan, Hubei
  - tongji Medical University, Wuhan, Hubei
  - Wuhan general hospital of Guangzhou command, Wuhan,chongqing, Hubei